CLINICAL TRIAL: NCT03958305
Title: An International European Retrospective Cohort Observational Study Comparing Laparoscopic or Robotic Radical Hysterectomy Versus Abdominal Radical Hysterectomy in Patients With Stage IB1 (FIGO 2009) Cervical Cancer Operated in 2013-2014
Brief Title: SUCCOR-Surgery in Cervical Cancer Comparing Different Surgical Aproaches in Stage IB1 Cervical Cancer
Acronym: SUCCOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: SUCCOR
Record Dates: First submitted 2019-04-15; First posted 2019-05-22 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-04

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LAPAROTOMY: Radical hysterectomy by laparotomy
  Interventions: Procedure: RADICAL HYSTERECTOMY
- MINIMALLY INVASIVE SURGERY: Radical hysterectomy by minimally invasive surgery (Laparoscopy or Robotics)
  Interventions: Procedure: RADICAL HYSTERECTOMY

INTERVENTIONS:
Procedure: RADICAL HYSTERECTOMY — Radical hysterectomy is an operation done to treat some cancers of the cervix. The surgeon takes out the uterus and the ligaments (tissue fibers) that hold it in place. The cervix and an inch or 2 of the vagina around the cervix are also removed.

SUMMARY:
SUCCOR study tries to understand the outcomes of European patients with stage IB1 cervical cancer (FIGO 2009)1, that underwent a radical hysterectomy for cervical cancer in 2013-2014 within the ESGO area (European Society of Gynecologic Oncology)

DETAILED DESCRIPTION:
SUCCOR study tries to understand the outcomes of European patients with stage IB1 cervical cancer (FIGO 2009) (1), that underwent a radical hysterectomy for cervical cancer in 2013-2014 within the ESGO area.

1.-Pecorelli, S. Revised FIGO staging for carcinoma of the vulva, cervix, and endometrium. Int J Gynaecol Obstet 105, 103-104 (2009).

Investigators want to know if the different surgical approaches may influence patients' survival (DFI and OS). A recent randomized phase III clinical trial, the LACC trial, conducted by Dr. Pedro Ramirez, was recently published in the NEJM.https://www.nejm.org/doi/pdf/10.1056/NEJMoa1806395

The LACC trial ran at 33 centers in 12 countries, including six US centers. The study, randomized women during 2008-2017 who had stage 1A1, 1A2, or 1B1 cervical cancer to either MIS or open surgery for a radical hysterectomy. The study's primary endpoint was disease-free survival at 4.5 years. The results favored significantly open surgery.

Just after this report, the results from a second study by Dr. Jose Alejandro Rauh-Hain, that used observational data from the US National Cancer Database found significantly worse overall survival following minimally invasive radical hysterectomy for early-stage cervical cancer, compared with laparotomy.

Also, Dr. Daniel Jacob Margul et al. presented during the last ASCO meeting their results from the Premier Health Database and the US National Cancer Database showing among women with >2 cm stage IB1 cervical cancer that MIS was associated with significantly decreased survival.

Likewise, these two studies have been as well published together along with the LACC trial in the same issue of NEJM.

In a recent survey conducted by the investigators and supported by ESGO, many of respondents showed the determination of collaborating in this observational project.

In Europe, it has not been recently not carried out any relevant large study comparing the different forms of surgical treatment of early cervical cancer.

The design of a randomized clinical trial in the coming years on this subject will face severe difficulties to convince ethics committees after the results of the last clinical trial.

Therefore, in the meantime, investigators consider it crucial to carry out a highly controlled European retrospective study that allows drawing satisfactory conclusions to make rational decisions on the treatment of early cervical cancer.

Investigators have selected a thorough list of inclusion and exclusion criteria along with a precise questionnaire trying to avoid confounding variables.

As you will realize, we will only include patients stage IB1(<4 cm, FIGO 2009), with preoperative MRI and with some requirements on the pathological report. For instance, patients that underwent conization are excluded.

HOW TO PARTICIPATE

1. Only centers belonging to the ESGO area can participate in the study
2. To accept the participation in the study as principal investigator (PI) of your institution (only one PI by each institution), the participant has to fill the application form included in the following link https://forms.gle/2WPhzrkxyFPodmDq5
3. As soon a center joins the study, the local PI will receive a Center Identification code and e-mail with instructions, allowing the data collection.
4. PI the will be allowed starting to collect data of consecutive cervical cancer patients operated in 2013 and 2014 in your center that meet the inclusion and exclusion criteria. (Appendix 2).
5. For collecting data, the online questionnaire can be reached in the following link: https://forms.gle/H1hCqXoC7G2EdWc79
6. Every time submit each a complete form, you will receive an e-mail with the confirmation and a copy of your response. For sending the form, you have to fill at least the required items. You are allowed to re-edit your answers later.
7. Investigators want to complete the data collection in less than six months.
8. The principal investigator will be available for any doubt by e-mail (lchiva@unav.es), or also by phone (+34630232947)
9. Besides, all the support documents will be sent to participants

PUBLICATIONS

The results of this study will be submitted for evaluation to international meetings and publication in a relevant international journal.

Authorship will include investigators following strict criteria, considering the introduced number of cases in the study by each investigator.

Furthermore, to count with as many authors as possible, researchers will create a Succor Research Study Group that will offer authorship when the investigators cannot allocate among the first authors

At the time of the publication, we will follow the STROBE guidelines for observational studies. (2) STROBE stands for an international, collaborative initiative of epidemiologists, methodologists, statisticians, researchers and journal editors involved in the conduct and dissemination of observational studies, with the common aim of STrengthening the Reporting of OBservational studies in Epidemiology.

(2) von Elm E, Altman DG, Egger M, Pocock SJ, Gøtzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE)statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9.

SUMMARY

The primary goal of the study is to know the outcomes of European patients that underwent radical surgery for stage IB1 cervical cancer (Open vs. MIS) during years 2013 and 2014.

ELIGIBILITY:
Inclusion criteria

* Primary squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix
* Stage IB1 carcinoma, <4 CMS, (FIGO 2009)
* Preoperative pelvic MRI indicating tumor diameter < 4 cm (at least two dimensions,) and no parametrial invasion. Exceptionally it can be considered acceptable Vaginal Ultrasound, only if your Institution have internally validated this technique for cervical cancer. Otherwise it cannot be accepted.
* Preoperative either (Abdominal) CT scan or MRI or PET-CT ruling out extracervical metastatic disease
* Performance status ECOG 0-1
* Age 18 years or older
* Radical hysterectomy Type II-III or Type B-C by MIS (laparoscopic or robotic) or open surgery.
* Patient was operated during the years 2013-2014 within the ESGO area.
* Bilateral pelvic lymphadenectomy (+- sentinel LN biopsy)
* Pathologic report shows information on tumor size, vaginal and parametrial margins and nodal status

Exclusion criteria

* No past medical history of any invasive tumor
* No previous abdominal or pelvic radiotherapy of any type (including braquitherapy).
* No history of preoperative neoadjuvant chemotherapy .
* No cervical conization previous to surgery
* No suspicious positive pelvic or paraaortic nodes or metastatic disease on PET CT, MRI, or CT.
* There is none uterine diameter larger than 12cm
* No Conversion from MIS to laparotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive participant sampling of patients with IB1 cervical cancer that underwent a Radical Hysterectomy plus pelvic lymphadenectomy by open or MIS
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival at 4.5 years | From date of surgery for cervical cancer (Radical Hysterectomy) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 84 months
  Compare disease-free survival at 4.5 years in patients who underwent a laparoscopic or robotic radical hysterectomy (MIS) vs. abdominal radical hysterectomy (TARH) for stage IB1 cervical cancer.

SECONDARY OUTCOMES:
Overall survival Overall survival at 5 years between groups. | months until the date of first documented date of death from any cause or the date last contact if case patient is alive, assessed up to 84 months
  Compare overall survival at 5 years in patients who underwent a laparoscopic or robotic radical hysterectomy (MIS) vs. abdominal radical hysterectomy (TARH) for stage IB1 cervical cancer.
Patterns of recurrence | Through study completion, an average of 1 year
  Compare patterns of recurrence between groups.
Rate of surgical complications during the first 30 days after surgery | 30 days after surgery
  Compare treatment-associated morbidity (30 days after surgery ) between groups

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Chiva, MD, PhD, Study Chair — Clinica Universidad de Navarra; Luis M Chiva, MD, PhD, Study Director — Clinica Universidad de Navarra; Daniel Vazquez, MD, PhD, Principal Investigator — Clinica Universidad de Navarra; Jose A Minguez, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: Yes
It will be uploaded in the network and it will be reached by a link provided by the promotors
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: January 2020
Access Criteria: It will be necessary to send an official request to the promotors

REFERENCES:
- [Background] Ramirez PT, Frumovitz M, Pareja R, Lopez A, Vieira M, Ribeiro R, Buda A, Yan X, Shuzhong Y, Chetty N, Isla D, Tamura M, Zhu T, Robledo KP, Gebski V, Asher R, Behan V, Nicklin JL, Coleman RL, Obermair A. Minimally Invasive versus Abdominal Radical Hysterectomy for Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1895-1904. doi: 10.1056/NEJMoa1806395. Epub 2018 Oct 31. PMID 30380365